CLINICAL TRIAL: NCT02110966
Title: Efficacy of the Combination Mepivacaine-Tramadol on the Success of Inferior Alveolar Nerve Block in Patients With Symptomatic Irreversible Pulpitis: a Randomized Clinical Trial.
Brief Title: Mepivacaine-Tramadol on the Success of Inferior Alveolar Nerve Block in Symptomatic Irreversible Pulpitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Daniel Chavarría Bolaños (Other)
Responsible Party: Sponsor-Investigator, Daniel Chavarría Bolaños, Basic Sciences Laboratory, Dentistry School, Universidad Autonoma de San Luis Potosí
Organization: Universidad Autonoma de San Luis Potosí (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIFE-008-014
Record Dates: First submitted 2014-04-08; First posted 2014-04-10 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Symptomatic Irreversible Pulpitis
Keywords: Anaesthetic effect; Inferior alveolar nerve block; Local tramadol; Mepivacaine; Symptomatic irreversible pulpitis.
MeSH Terms: interventions — Mepivacaine; Tramadol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mepivacaine plus Tramadol (Experimental): 1.3 ml of Mepivacaine 2% epinephrine 1:100000 mixed with 0.5 ml of Tramadol (50mg/ml) will be used for the anesthetic blockade in the experimental group
  Interventions: Drug: Mepivacaine plus Tramadol
- Mepivacaine (Active Comparator): The control group will receive the inferior alveolar nerve block using 1.8 ml of Mepivacaine 2% epinephrine 1: 100000.
  Interventions: Drug: Mepivacaine

INTERVENTIONS:
Drug: Mepivacaine — Drug: Tramadol 1.8 ml of Mepivacaine 2% epinephrine 1:100000.
  Other Names: Dentocaín
  Arms: Mepivacaine
Drug: Mepivacaine plus Tramadol — 0.5 ml of Tramadol mixed with 1.3 ml of Mepivacaine.
  Other Names: Tradol
  Arms: Mepivacaine plus Tramadol

SUMMARY:
The purpose of this study is to evaluate the success of inferior alveolar nerve block, after the local application of Mepivacaine plus Tramadol in patients with symptomatic irreversible pulpitis. Also, to evaluate the duration of the anesthetic effect when using Mepivacaine plus Tramadol in the same anesthetic technique and patients group.

Hypothesis:

Local application of mepivacaine plus tramadol increases the successful of inferior alveolar nerve block in patients with irreversible pulpitis.

DETAILED DESCRIPTION:
The treatment of pain is an integral part of Endodontics, this must be controlled before, during and after treatment. The inferior alveolar nerve block is the most common anesthetic technique used in mandibular teeth during endodontic treatments. Several studies have reported that it is more difficult to obtain anesthetic success in patients with irreversible pulpitis. There is a 33-80% of failure in the inferior alveolar nerve block in patients with irreversible pulpitis.

Some of the more accepted theories for local anesthetic failure establish that inflammation induce tissue acidosis causing ion traping of the local anesthetics enabling the molecules to cross the cell membrane, also inflammatory mediators may sensitize the neurons by interacting with specific receptors leading to periphery sensibilization. Tissue injury may alter the composition, distribution and activity of sodium channels expressed on nociceptors and this may have profound implications in local anesthetic failure. On the other hand, there is a specific group of tetrodotoxin resistant sodium channels four times less sensitive to lidocaine which increase their activity during inflammation.

Some ways to control pain is through pharmacological synergism. Tramadol has been proposed as pharmacological adjuvant to local anesthesia and it can improve the anesthetics success and the duration of the anesthetic effect. However, oral administration of drugs can cause adverse systemic effects, and that's why local application is an alternative to increase its concentration on the local damaged tissue reducing the possibility of interactions with other drugs and adverse effects. Another advantage of the combination of Mepivacaine with Tramadol is that it reduces the number of injections in patients and it is less traumatic.

Tramadol is centrally acting drug but also a local anesthetic and analgesic effect it has been reported. It acts at multiple sites producing different action mechanisms. Some studies suggest that the use of Tramadol can improve the effect of Mepivacaine in the inferior alveolar nerve block. The blockade of the nervous conduction with Tramadol is 80% more effective if it is compared with some anesthetics like lidocaine.

There are few studies evaluating local application of tramadol. In the field of dentistry tramadol using for local anesthetic adjuvant has been studied in oral surgery, so it is important to evaluate it in the field of endodontics to provide better pain management during treatments.

Thus, the aim of the study is to evaluate the success of inferior alveolar nerve block with the local application of Mepivacaine plus Tramadol in patients with symptomatic irreversible pulpitis, and also to evaluate the duration of the anesthetic effect when using Mepivacaine plus Tramadol in the anesthetic technique. This study was designed as a double-blind, randomized clinical trial. Following the guidelines suggested by CONSORT group for planning and reporting clinical trials. The ethics committee of the Faculty of Dentistry of San Luis Potosi University approved the study design. All of the subjects will be informed of the possible risk of endodontic therapy and experimental treatments and will sign institutionally approved consents forms.

In total 50 patients will be included in this study. The sample size calculation was performed with a Type I error of 0.05 and statical power of 80% using the difference in duration of anesthetic effect between two groups and taking into account previous studies related to the local effect of tramadol in clinical studies where it is used to assess the time of anesthetic effect.

All the subjects voluntarily will presented at the Postgraduate Endodontics Clinic of the Faculty of Dentistry at San Luis Potosi University. The select subjects will have a diagnosis of symptomatic irreversible pulpitis in the first and second mandibular molars.

The patients will be diagnosing with the cold test and they will indicate their pain scores using numerical rating scale, this is a 11 point scale where the ends points are the extremes of no pain and the worst pain. Accordingly, no pain corresponded with 0, mild pain with 1-3, moderate pain with 4-6 and severe pain 7-10. The control group will receive the inferior alveolar nerve block using 1.8 ml of Mepivacaine 2% epinephrine 1: 100000 and 1.3 ml of Mepivacaine 2% epinephrine 1:100000 mixed with 0.5 ml of Tramadol (50mg/ml) will be used for the anaesthetic blockade in the experimental group. After 15 minutes, the anesthetic blockade will be assessed by a three step examination: lip numbess, positive/negative response to cold testing and clinical discomfort during endodontic access. Inferior alveolar nerve block success will be defined as the absence of pain during any of these evaluations and if patients report pain an analogue visual scale will be used.

Statics normal distribution will be tested by the student's t test. A non-parametric chi- squared test was performed to identify statistically differences between the groups; the level of significance was set at p˂ 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with symptomatic irreversible pulpitis in the first and second mandibular molars.

Exclusion Criteria:

* Pregnancy
* Hypersensitivity to local anesthetics and Tramadol
* Teeth with insufficient tooth structure for restoration, periodontal disease, root resorption, root fracture
* Systemic diseases: diabetes, uncontrolled hypertension.
* Patients taking drugs or narcotics.
* Patients who have used analgesics in the last 8 hours.
* Patients ingested IMAOS and tricyclic antidepressants 14 days before.
* Patients ingested carbamazepine (anticonvulsants)
* Patients in active treatment with ketoconazole and erythromycin.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
success of the inferior alveolar nerve block | 0-30 minutes
  The anesthetic blockade will be assessed by a three step examination: lip numbess, positive/negative response to cold testing and clinical discomfort during endodontic access. Inferior alveolar nerve block success will be defined as the absence of pain during any of these evaluations and if patients report pain an analogue visual scale will be used. Also, the patient will reported the level of pain in the application of the inferior alveolar nerve block using mepivacaine and mepivacaine plus tramadol and local and systemic side effects will be monitored.

SECONDARY OUTCOMES:
Anesthetic effect duration | 0-14 hours
  The time of the anesthetic effect will be evaluated in patients in whom anesthetic success is achieved, and also the consume of emergency and rescue post-operative analgesics. Side effects will also be monitored during this period.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Rodríguez, DDS, Principal Investigator — Universidad Autónoma San Luis Potosí; Daniel Chavarria, MSc, PhD, Study Director — Universidad Autonoma San Luis Potosi; Amaury Pozos, MSc, PhD, Study Chair — Universidad Autonoma San Luis Potosi
Locations (1):
- Endodontics Master Degree program, Dentistry Faculty, San Luis Potosi University, San Luis Potosí City, San Luis Potosí, Mexico

REFERENCES:
- [Background] Walton RE, Torabinejad M. Managing local anesthesia problems in the endodontic patient. J Am Dent Assoc. 1992 May;123(5):97-102. doi: 10.14219/jada.archive.1992.0133. PMID 1597649
- [Background] Hellstrom PM, Husebye E, Kraglund K. Methodology for motility studies on the small intestine: a Scandinavian consensus. Eur J Surg Suppl. 1991;(564):51-61. No abstract available. PMID 1718505
- [Background] Cohen HP, Cha BY, Spangberg LS. Endodontic anesthesia in mandibular molars: a clinical study. J Endod. 1993 Jul;19(7):370-3. doi: 10.1016/S0099-2399(06)81366-X. PMID 8245762
- [Background] Henry MA, Hargreaves KM. Peripheral mechanisms of odontogenic pain. Dent Clin North Am. 2007 Jan;51(1):19-44, v. doi: 10.1016/j.cden.2006.09.007. PMID 17185058
- [Background] Noguera-Gonzalez D, Cerda-Cristerna BI, Chavarria-Bolanos D, Flores-Reyes H, Pozos-Guillen A. Efficacy of preoperative ibuprofen on the success of inferior alveolar nerve block in patients with symptomatic irreversible pulpitis: a randomized clinical trial. Int Endod J. 2013 Nov;46(11):1056-62. doi: 10.1111/iej.12099. Epub 2013 Apr 6. PMID 23561002
- [Background] Kargi E, Babuccu O, Altunkaya H, Hosnuter M, Ozer Y, Babuccu B, Payasli C. Tramadol as a local anaesthetic in tendon repair surgery of the hand. J Int Med Res. 2008 Sep-Oct;36(5):971-8. doi: 10.1177/147323000803600513. PMID 18831890
- [Background] Sawynok J. Topical and peripherally acting analgesics. Pharmacol Rev. 2003 Mar;55(1):1-20. doi: 10.1124/pr.55.1.1. PMID 12615951
- [Background] Stein C, Lang LJ. Peripheral mechanisms of opioid analgesia. Curr Opin Pharmacol. 2009 Feb;9(1):3-8. doi: 10.1016/j.coph.2008.12.009. Epub 2009 Jan 20. PMID 19157985
- [Result] Isiordia-Espinoza MA, Pozos-Guillen AJ, Martinez-Rider R, Herrera-Abarca JE, Perez-Urizar J. Preemptive analgesic effectiveness of oral ketorolac plus local tramadol after impacted mandibular third molar surgery. Med Oral Patol Oral Cir Bucal. 2011 Sep 1;16(6):e776-80. doi: 10.4317/medoral.16854. PMID 21217614
- [Result] Wang JT, Chung CC, Whitehead RA, Schwarz SK, Ries CR, MacLeod BA. Effects of local tramadol administration on peripheral glutamate-induced nociceptive behaviour in mice. Can J Anaesth. 2010 Jul;57(7):659-63. doi: 10.1007/s12630-010-9301-9. Epub 2010 Mar 26. PMID 20340056
- [Result] Robaux S, Blunt C, Viel E, Cuvillon P, Nouguier P, Dautel G, Boileau S, Girard F, Bouaziz H. Tramadol added to 1.5% mepivacaine for axillary brachial plexus block improves postoperative analgesia dose-dependently. Anesth Analg. 2004 Apr;98(4):1172-1177. doi: 10.1213/01.ANE.0000108966.84797.72. PMID 15041620
- [Result] Guven M, Mert T, Gunay I. Effects of tramadol on nerve action potentials in rat: comparisons with benzocaine and lidocaine. Int J Neurosci. 2005 Mar;115(3):339-49. doi: 10.1080/00207450590520948. PMID 15804720
- [Result] Isiordia-Espinoza MA, Orozco-Solis M, Tobias-Azua FJ, Mendez-Gutierrez EP. Submucous tramadol increases the anesthetic efficacy of mepivacaine with epinephrine in inferior alveolar nerve block. Br J Oral Maxillofac Surg. 2012 Mar;50(2):157-60. doi: 10.1016/j.bjoms.2011.02.010. Epub 2011 May 8. PMID 21555171
- [Result] Altunkaya H, Ozer Y, Kargi E, Ozkocak I, Hosnuter M, Demirel CB, Babuccu O. The postoperative analgesic effect of tramadol when used as subcutaneous local anesthetic. Anesth Analg. 2004 Nov;99(5):1461-1464. doi: 10.1213/01.ANE.0000135640.21229.A0. PMID 15502049
- [Result] Pozos AJ, Martinez R, Aguirre P, Perez J. The effects of tramadol added to articaine on anesthesia duration. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2006 Nov;102(5):614-7. doi: 10.1016/j.tripleo.2006.01.017. Epub 2006 Jul 27. PMID 17052637
- [Result] Kapral S, Gollmann G, Waltl B, Likar R, Sladen RN, Weinstabl C, Lehofer F. Tramadol added to mepivacaine prolongs the duration of an axillary brachial plexus blockade. Anesth Analg. 1999 Apr;88(4):853-6. doi: 10.1097/00000539-199904000-00032. PMID 10195537
- [Result] Ceccheti MM, Negrato GV, Peres MP, Deboni MC, Naclerio-Homem Mda G. Analgesic and adjuvant anesthetic effect of submucosal tramadol after mandibular third molar surgery. Oral Surg Oral Med Oral Pathol Oral Radiol. 2014 Mar;117(3):e249-54. doi: 10.1016/j.oooo.2012.05.015. Epub 2012 Sep 12. PMID 22981094
- [Result] Pozos AJ, Martinez R, Aguirre P, Perez J. Tramadol administered in a combination of routes for reducing pain after removal of an impacted mandibular third molar. J Oral Maxillofac Surg. 2007 Aug;65(8):1633-9. doi: 10.1016/j.joms.2006.06.267. No abstract available. PMID 17656294